CLINICAL TRIAL: NCT05276089
Title: Evaluating the Impact of an Evidence Informed, Digitally Deployed, GP Remote Consultation Video Intervention That Aims to Reduce Opioid Prescribing in Primary Care
Brief Title: GP Remote Consultation to Reduce Opioid Prescribing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Yu Fu (Other)
Collaborators: Teesside University (Other); NIHR Applied Research Collaboration for North East and North Cumbria (Unknown); North East Academic Health Science Network (Unknown)
Responsible Party: Sponsor-Investigator, Dr Yu Fu, Principal Investigator, Newcastle University
Organization: Newcastle University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NU-010572
Record Dates: First submitted 2022-02-21; First posted 2022-03-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): A total of 50 practices who use System 1 will be in the intervention arm to send out the video to their eligible patients.
  Interventions: Behavioral: Video message
- Control arm (No Intervention): 50 practices who use EMIS will be in the control arm to deliver care as usual

INTERVENTIONS:
Behavioral: Video message — The five-minute video will be sent to the patient's mobile phone, outlining reasons to reduce opioid use and highlighting the support available. It invites patients to consider 3 responses:
  1. I would like to reduce my opioid medication with support.
  2. I understand this video but I want to continue my current dose.
  3. I would like to speak to someone to understand more. Option 1) will enable the GP practice to initiate existing opioid reduction support, Option 2) will continue care and support as usual, and Option 3) will enable the team to offer more information.
  Arms: Intervention arm

SUMMARY:
Opioid prescribing rates are high in the North East and North Cumbria region of England. The COVID-19 pandemic has interrupted the existing regional programme that aims to reduce the use of opioid medications, and also prescribing is likely to have increased during the lockdown. Thus, it has become increasingly challenging for primary care to dedicate sustained clinical time to tackle this complex issue with patients, who may also be reluctant to seek help. A video messaging intervention based upon a GP consultation was developed to remotely explain the rationale for opioid reduction and facilitate self-initiation of support. The short video suitable for smartphone viewing is messaged using a two-way communication system. Patients can watch the video and request additional support by replying with a simple text or email response. This enables efficient delivery of a discrete offer of help to at risk individuals who often avoid service contact. The aim of this study is to evaluate the potential benefits, risks and economic consequences of 'at scale' implementation.

This study will be a mixed methods study comprising of a quasi-experimental non-randomised before-and-after study and qualitative interviews. In the first phase, the intervention arm will comprise 50 GP practices in the region using System 1 who will deliver the video to their patients. The control arm comprises 50 practices in the region using EMIS who will continue care as usual. The unit of analysis is the GP practice, with no individual-level quantitative data collected. Monthly practice level data will be accessed and followed up for 6 months. A general linear model will be used to estimate the association between the exposure (video message vs. control) and the outcome (opioid prescribing). In the second phase, semi-structured interviews will be undertaken remotely with purposively selected participants including patients who received the video and health professionals involved in sending out the videos. These interviews will be audio recorded with participants' consent, transcribed and analysed thematically.

As well as evidence and rapid insights to inform the potential accelerated implementation of the intervention within the Integrated Care System, this study will provide evidence that could underpin the future adoption of the intervention into wide scale clinical management that can be disseminated as a future national programme via the Academic Health Science Network.

ELIGIBILITY:
Inclusion Criteria:

* adults (aged 18 or over)
* registered with a mobile phone number at practices
* regularly taking opioids for more than 90 days or at a dose equivalent to > 100 mg of codeine a day (this varies for each opioid medication) using electronic records

Exclusion Criteria:

* if they are coded cancer or palliative care.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline line opioids analgesics assessed as Average Daily Quantity (ADQ)/1000 Specific Therapeutic group Age-sex Related Prescribing Unit (STAR PU) at 6 months | Up to 7 months
  This is a practice level data collected monthly by electronic Prescribing Analysis and Costs (ePACT2) by North of England Commissioning Support Unit (NECS). NECS has agreed to support data requests and access.

SECONDARY OUTCOMES:
Change from baseline line all opioids (adding in compound analgesics) Average Daily Quantity (ADQ)/1000 Specific Therapeutic group Age-sex Related Prescribing Unit (STAR PU)at 6 months | Up to 7 months
  This is a practice level data collected monthly by electronic Prescribing Analysis and Costs (ePACT2) by North of England Commissioning Support Unit (NECS). NECS has agreed to support data requests and access.
Change from baseline line gabapentinoid (gabapentin&pregabalin) Average Daily Quantity (ADQ)/1000 Specific Therapeutic group Age-sex Related Prescribing Unit (STAR PU) at 6 months | Up to 7 months
  This is a practice level data collected monthly by electronic Prescribing Analysis and Costs (ePACT2) by North of England Commissioning Support Unit (NECS). NECS has agreed to support data requests and access.
Change from baseline line high dose opioid items as percentage regular opioids | Up to 7 months
  Information on high dose opioid items as percentage regular opioids will be collected from the publicly accessible dataset (OpenPrescribing.net), which records monthly data on opioid items with likely daily dose of ≥120mg morphine equivalence compared with prescribing of all items of these opioids.
The number (proportion) of individuals who were followed up by the practice within 1 month of choosing Options 1) and 3), will be quantified being sent the message. | Up to 7 months
  Intervention usage
The percentage of the video watched by participants who were sent the video | Up to 7 months
  Fidelity
Intervention costs | Up to 7 months
  Intervention costs will be estimated based on interviews with the developer of the videos and GP practice stakeholders to understand the licence costs and the opportunity costs of practice staff time in finding the appropriate population to whom the videos will be sent. If applicable, the investigators will estimate any additional resources needed by people receiving videos who decide to reduce or eliminate their opioid use, who may need GP practice visits to discuss this.

CONTACTS AND LOCATIONS:
Locations (1):
- LCRN, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no IPD involved in this trial.

REFERENCES:
- [Derived] Fu Y, Allen B, Batterham AM, Price C, Jones N, Martin D, Hex N, Maule E, Finch T, Newton JL, Ryan CG. Digitally deployed, GP remote consultation video intervention that aims to reduce opioid prescribing in primary care: protocol for a mixed-methods evaluation. BMJ Open. 2023 Feb 6;13(2):e066158. doi: 10.1136/bmjopen-2022-066158. PMID 36746541